CLINICAL TRIAL: NCT06226818
Title: Assessing the Impact on Mental and Physical Health of Caring for Women Who Are Victims of Sexual and Gender-based Violence, Using a Coordinated Multidisciplinary Approach in Women's or Traditional Health Centres: a Prospective, Quasi-experimental, Multicentre, National Study.
Brief Title: Evaluation of the Impact on Mental and Physical Health of Caring for Women Who Are Victims of Sexual and Gender-based Violence, Using a Coordinated Multidisciplinary Approach in Women's Centres or Traditional Health Centres.
Acronym: IROND-L
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BARDOU PREPS 2022
Record Dates: First submitted 2024-01-18; First posted 2024-01-26 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Domestic and/or Sexual Violence
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- experimental group: Women cared for in a women's centre
  Interventions: Other: completion of scales and questionnaires
- comparator group: Women in a health centre or family planning centre.
  Interventions: Other: completion of scales and questionnaires

INTERVENTIONS:
Other: completion of scales and questionnaires — Patient questionnaires Abuse assessment Screen, Evaluation of the PCL-5 score, Measurement of insomnia severity indexes (ISI), quality of life scores (WHOQOL-BREF), anxiety and depression using the HAD scale (Hospital Anxiety and Depression), self-esteem score using the Rosenberg scale, feeling of security and well-being using five-point Likert scales.
  Questionnaire on daily and occasional smoking, alcohol consumption using the Alcohol Use Disorders Identification Test-Concise (AUDIT-C), cannabis dependence using the Cannabis Abuse Screening Test (CAST) and use of other psychoactive substances.

SUMMARY:
Gender-based or sexual violence, or violence against women (VAW), is a global public health problem affecting around 30% of women over the age of 15, with significant consequences for physical and mental health, including depression and post-traumatic stress disorder (PTSD).

In 2019, the French National Authority for Health (HAS) published recommendations in two parts, one for identifying women who are victims of domestic violence, and the other for dealing with a woman who has been exposed to such violence. But violence against women is not limited to the marital sphere. VAW can simply be detected in a consultation using a translated version of the Abuse Assessment Screen (AAS) questionnaire.

Women who are victims of VAW have specific needs linked to the often repeated nature of the violence they experience, and the complex trauma that can ensue. They also tend to combine other risk factors for poor mental health, such as economic insecurity and social isolation. In France, dealing with the specific medical, psychosocial and legal needs of victims-survivors of VAW has come up against a number of obstacles, including a lack of dedicated care facilities, a lack of trained professionals and a lack of coordination between the various parties. Health professionals rarely receive the training they need to deal with VAW-related issues with confidence and professionalism, and often lack the resources to refer female victims to appropriate care.

"La Maison des Femmes" (MdF) was set up in 2016 in Saint-Denis, located in a department where a quarter of the women who consult a family planning centre (FPC) has suffered from VAW. It is a hospital service specifically dedicated to the individualised, multidisciplinary care of victims-survivors of VAW, offering health, social and legal support within the same facility. The MdF comprises 4 units: a FPC, a violence management unit (involving doctors, midwives, psychologists, social workers, lawyers, police officers and support groups), a female genital mutilation management unit (surgeons and sexologists) and a 24/7 reception unit for victims of sexual violence.

Several MdF-inspired care structures have been set up in France. The service provided by these facilities needs to be evaluated, particularly in terms of their ability to improve the physical and mental health, including post-traumatic stress, of women who have been victims of VAW.

ELIGIBILITY:
Inclusion Criteria:

* Women who have not objected to taking part in the trial
* Adult women (≥18 years),
* Victim of domestic and/or sexual violence, consulting at one of our study centres. Exposure to violence, whatever the initial reason for consultation, will be determined by a positive response to at least one question on the French version of the Abuse Assessment Screen, a standardised screening tool which has the advantage of not being limited to domestic violence.
* Ability to understand the objectives of the study and to answer the questionnaires

Exclusion Criteria:

* Not affiliated to the national health insurance system
* Person under legal protection (curatorship, guardianship)
* Person under court order
* Adult who is unable to express his/her non-opposition
* Minor

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients will be identified by a doctor at one of the participating centres, on the basis of their response to the AAS questionnaire during the initial consultation.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2024-08-08 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Change in mean PCL-5 score | Through study completion, an average of 6 months
  measured using the validated French version of the Post-traumatic Stress Disorder Checklist for DSM-V (score from 0 to 80).
Change in the proportion of women with a PCL-5 score < 33 (validated threshold for absence of overt PTSD) | Through study completion, an average of 6 months
  measured using the validated French version of the Post-traumatic Stress Disorder Checklist for DSM-V (score from 0 to 80).

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Khoury F, Ben Ghezala I, Hatem G, Jaffal Z, Soares A, Yacini L, Duchesne S, Dommergues M, Bretelle F, Eudeline S, Hoffmann P, Masse-Navette C, Layachi F, Maurice O, de Foucher de Careil T, Bardou M. IROND-L: study protocol for a French prospective, quasi-experimental, multicentre trial to examine the impact of a coordinated multidisciplinary approach for women victims of violence. BMJ Open. 2024 Nov 19;14(11):e086143. doi: 10.1136/bmjopen-2024-086143. PMID 39566954